CLINICAL TRIAL: NCT06409507
Title: The Impact of FKBP12 on the Prognosis and Sirolimus Administration in Liver Transplantation Recipients With Hepatocellular Carcinoma: A Single-center Retrospective Cohort Study
Brief Title: Research and Application for New Clinical Diagnosis and Treatment System for HBV Related HCC Liver Transplantation
Status: Completed | Type: Observational
Sponsor: First People's Hospital of Hangzhou (Other)
Responsible Party: Sponsor
Other Study IDs: 2018768
Record Dates: First submitted 2024-05-07; First posted 2024-05-10 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-03

CONDITIONS: Hepatocellular Carcinoma; Liver Transplantation; Prognosis
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Sirolimus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- high FKBP12 expression: The immunoreactive score (IRS), calculated by multiplying the staining intensity grades by the proportion of positive cells, was used to assess the expression levels of FKBP12. IRS (8-12) represented high expression levels.
  Interventions: Genetic: FKBP12 expression
- low FKBP12 expression: The immunoreactive score (IRS), calculated by multiplying the staining intensity grades by the proportion of positive cells, was used to assess the expression levels of FKBP12. IRS (0-7) represented low expression levels.
  Interventions: Genetic: FKBP12 expression

INTERVENTIONS:
Genetic: FKBP12 expression — The expressions of FKBP12 were determined by immunohistochemistry (IHC) , and the immunoreactive score (IRS), calculated by multiplying the staining intensity grades by the proportion of positive cells, was used to assess the expression levels of FKBP12. IRS (0-7) represented low expression levels, and IRS (8-12) represented high expression levels.
  Other Names: sirolimus

SUMMARY:
The study evaluated the protein expression levels of FK506-binding protein 12 (FKBP12) in hepatocellular carcinoma (HCC) and paracancerous tissues using immunohistochemistry (IHC). This study aimed to determine the role of FKBP12 in the outcome of liver transplantation recipients with HCC, especially those exceeding the Milan criteria. In addition, we explored how sirolimus administration affected LT recipients'prognosis depending on different FKBP12 expression, aiming to provide some advice for clinical sirolimus application after LT.

ELIGIBILITY:
Inclusion Criteria:

* (1) pathologically confirmed HCC (2) full post-LT follow-up record

Exclusion Criteria:

* (1)sirolimus treatment less than 30 days or after tumor recurrence (2)died within 90 days (3)underwent multiple-organ transplantation

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Deceased donor LT surgery was performed in all recipients at our center between January 1, 2015 and January 1, 2021. China Liver Transplant Registry database (http://www.cltr.org) was used to obtain clinical information about patients, which included age, gender, pathological characteristics, pre-LT alpha-fetoprotein (AFP), loco-regional therapy (including transcatheter arterial chemoembolization (TACE) and radiofrequency ablation (RFA)) before LT, model for end-stage liver disease (MELD) score, Child-Pugh score, hepatitis B virus status, sirolimus administration, date of surgery, recurrence, last follow up, and death. LT recipients were required for a follow-up examination every 3 months.
Sampling Method: Probability Sample
Enrollment: 178 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
Overall survival | 2015.1.1-2021.1.1
  the length of months between surgery and the last follow-up or death

IPD SHARING:
Plan to Share IPD: No